CLINICAL TRIAL: NCT02603601
Title: A Randomized Controlled Trial of Lifestyle Interventions to Control Weight After Bariatric Surgery
Brief Title: A Trial of Lifestyle Interventions to Control Weight After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Center for Nutritional Research Charitable Trust (Other)
Responsible Party: Principal Investigator, Christina Wee, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013P000259
Record Dates: First submitted 2015-02-04; First posted 2015-11-13 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Obesity; Weight Gain
Keywords: Randomized controlled trial; Mindfulness; Obesity
MeSH Terms: conditions — Obesity; Weight Gain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard lifestyle intervention (Active Comparator): The standard lifestyle intervention is a 1-hour individual nutritional counseling session with a registered dietician at BIDMC.
  Interventions: Behavioral: Standard lifestyle intervention
- Mind-body lifestyle intervention (Experimental): The mind-body lifestyle intervention is a 10-week mindfulness-based intervention that integrates mindfulness with traditional behavioral strategies to improve long-term weight maintenance.
  Interventions: Behavioral: Mind-body lifestyle intervention

INTERVENTIONS:
Behavioral: Mind-body lifestyle intervention
  Arms: Mind-body lifestyle intervention
Behavioral: Standard lifestyle intervention
  Arms: Standard lifestyle intervention

SUMMARY:
This randomized controlled trial is designed to test the feasibility and efficacy of a novel 10-week mindfulness-based intervention (MBI) on weight maintenance as well as behavioral and psychosocial outcomes in patients who have undergone bariatric surgery.

Primary hypothesis:

Bariatric patients who have stopped losing weight (< 5 lbs weight loss in past month) 1-5 years post-surgery will be willing to participate in this 10-week intervention. The investigators expect a high adherence rate (>70%) and no issues with meeting recruitment goals.

Secondary hypotheses:

Patients assigned to the MBI will show greater improvement in a) weight control (defined by differences in body weight between baseline and follow-up); b) eating behaviors (binge eating, emotional eating); and c) psychosocial measures (quality of life, depression, perceived stress, eating self-efficacy, coping ability) than a standard lifestyle intervention (1 hr lifestyle counseling).

Patients assigned to the MBI intervention will show greater improvement in biomarkers of stress and inflammation [salivary cortisol, high sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6), and tumor necrosis factor-alpha (TNF-alpha)] as compared with a standard lifestyle intervention.

Food-related attentional bias as measured by the food-related Stroop task will be differentially affected among patients assigned to the MBI as compared with the intensive lifestyle intervention and standard lifestyle intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have undergone bariatric surgery 1-5 years prior to study start (by medical record and/or self report)
2. Weight loss plateau (< 5 lbs weight loss in past month) (by medical report and/or self report)
3. Ages 18-65 years (by medical record and/or self report)
4. Able to complete outcome assessments

Exclusion Criteria:

1. Prior experience with meditation course (past 6 months), current mindfulness/meditation practice, or regular meditation or mindfulness practice in past year ("Regular practice" defined as practicing formally 1 or more times a week for 2 months).
2. Plans to leave the study area within next 12 months
3. Serious psychiatric illness or personality disorder (by medical record and/or self-report)
4. Current alcohol and/or substance abuse
5. Pregnancy or plans to become pregnant in next year
6. Non-English speaking
7. > 1 prior weight loss surgery (by medical record and self-report)
8. Gastric band removed prior to study contact.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Success meeting recruitment goals (20 patients within 3-4 months) | 4-month recruitment window
Willingness to participate in study (>10% of eligible) | 4-month recuitment window
Adherence rate (≥70% attendance, 7 of 10 classes) | 12-weeks
Retention (≤25% drop-out) | 6-months

SECONDARY OUTCOMES:
Changes in body weight as measured on a digital scale | 12 ± 2 weeks post intervention-baseline
Eating behaviors measured using the Three Factor Eating Questionnaire | 12 ± 2 weeks
Eating behaviors measured using the Binge Eating Scale | 12 ± 2 weeks
Quality of life measured using the Medical Outcomes Study Short-Form-36 scale | 12 ± 2 weeks
Quality of life measured using the Impact of Weight on Quality of Life scale | 12 ± 2 weeks
Depression measured by the Center for Epidemiologic Studies Depression Scale | 12 ± 2 weeks
Perceived stress measured by the Perceived Stress Scale | 12 ± 2 weeks
Ability to cope measured by the Brief Cope questionnaire | 12 ± 2 weeks
Eating self-efficacy measured by the Weight Efficacy Lifestyle Questionnaire | 12 ± 2 weeks

OTHER OUTCOMES:
Biomarkers of stress measured by bioassay techniques | 12 ± 2 weeks
Biomarkers of inflammation measured by bioassay techniques | 12 ± 2 weeks
Food-related attentional bias as measured by the Food-related Stroop task. | 12 ± 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christina C Wee, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconness Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Chacko SA, Yeh GY, Davis RB, Wee CC. A mindfulness-based intervention to control weight after bariatric surgery: Preliminary results from a randomized controlled pilot trial. Complement Ther Med. 2016 Oct;28:13-21. doi: 10.1016/j.ctim.2016.07.001. Epub 2016 Jul 12. PMID 27670865